CLINICAL TRIAL: NCT00471107
Title: Effect of Direct Current Brain Polarization on Verbal Memory
Brief Title: Effect of Electrical Stimulation (DC Polarization) to the Brain on Memory
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 070147; 07-N-0147
Record Dates: First submitted 2007-05-08; First posted 2007-05-09 (Estimated); Results first posted 2013-05-15 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Frontal Lobe; Language; Dementia; Healthy Volunteer; HV
MeSH Terms: conditions — Language; Dementia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sham TDCS (Sham Comparator)
  Interventions: Device: DC brain polarization
- Surface-anodal direct current (Experimental): 0.08 mA/cm2
  Interventions: Device: DC brain polarization
- Surface-cathodal direct current (Active Comparator): 0.08 mA/cm2
  Interventions: Device: DC brain polarization

INTERVENTIONS:
Device: DC brain polarization — 0.08 mA/cm2

SUMMARY:
This study will test the effect of direct current (DC) brain polarization (the application of a very weak electrical current to the brain) on learning and memory. Earlier studies have shown that DC polarization can temporarily improve the ability of healthy people to think of certain words. This study will explore whether it can also temporarily improve learning and memory.

Healthy people 18 years of age and older may be eligible for this study. Subjects participate in two experimental sessions at the NIH Clinical Center. The first session lasts about 1 hour; the second session, on the next day, takes about 10 minutes.

At the beginning of the first session, electrodes are placed on the subject's head and arm for brain stimulation. The current may be turned on for 25 minutes, or only very briefly (sham stimulation). Subjects are not told which type of stimulation they are receiving. No stimulation is applied in the second session.

During the sessions subjects are asked to complete the following tasks that will help elucidate the effects of polarization:

* Read a list of words and remember them. Later they will try to repeat the words from memory.
* Look at a series of designs and remember them. Later they will try to draw the designs from memory.
* Push a button on a keyboard when they see a specific item (for example, when the number 7 appears).
* Generate as many words as they can think of that begin with a particular letter of the alphabet.

Subjects may be videotaped for some or all of the time during the sessions.

DETAILED DESCRIPTION:
OBJECTIVE: The principal objective is to establish whether DC polarization of left lateral prefrontal cortex can enhance verbal memory.

STUDY POPULATION: 75 healthy volunteers over the age of 18 will be enrolled.

DESIGN: The study is a double-blind parallel study with three arms: anodal polarization, cathodal polarization, and sham treatment.

OUTCOME MEASURES: The primary outcome measure is performance on the WMS-III Word Lists test. Secondary outcome measures, testing for effects of DC polarization on basic information processing and non-verbal memory, respectively, are the CalCAP and WMS-III Visual Reproduction Test. The Verbal Fluency Test will be administered prior to stimulation and 24 hours post-stimulation to screen for other residual effects of the polarization on the stimulated region.

ELIGIBILITY:
* INCLUSION CRITERIA:

Healthy volunteers over age 18. Pregnancy is not an exclusion.

EXCLUSION CRITERIA:

Any history of a central nervous system illness or other behavioral disorder.

Broken skin in the area of the electrodes.

Uncontrolled medical problems, such as diabetes mellitus, hypertension, airway disease, heart failure, coronary artery disease, or any other condition that poses a risk for the subject during participation.

Presence of metal in the cranial cavity.

Holes in the skull made by trauma or surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2007-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Herwig U, Satrapi P, Schonfeldt-Lecuona C. Using the international 10-20 EEG system for positioning of transcranial magnetic stimulation. Brain Topogr. 2003 Winter;16(2):95-9. doi: 10.1023/b:brat.0000006333.93597.9d. PMID 14977202
- [Background] BINDMAN LJ, LIPPOLD OC, REDFEARN JW. Long-lasting changes in the level of the electrical activity of the cerebral cortex produced bypolarizing currents. Nature. 1962 Nov 10;196:584-5. doi: 10.1038/196584a0. No abstract available. PMID 13968314
- [Background] CREUTZFELDT OD, FROMM GH, KAPP H. Influence of transcortical d-c currents on cortical neuronal activity. Exp Neurol. 1962 Jun;5:436-52. doi: 10.1016/0014-4886(62)90056-0. No abstract available. PMID 13882165

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy subjects were recruited through the NIH Clinical Research Volunteer Program
Pre-assignment Details: Nothing to report
Groups:
- Anodal TDCS: Randomly selected healthy volunteers undergoing left dorsolateral prefrontal cortex (LDPFC) anodal transcranial direct current stimulation (tDCS) during verbal memory tasks.
- Cathodal TDCS: Randomly selected healthy volunteers undergoing left dorsolateral prefrontal cortex (LDPFC) cathodal transcranial direct current stimulation (tDCS) during verbal memory tasks.
- Sham TDCS: Randomly selected healthy volunteers undergoing left dorsolateral prefrontal cortex (LDPFC) sham stimulation during verbal memory tasks.
Period: Overall Study
Arm/Group | Anodal TDCS | Cathodal TDCS | Sham TDCS
Started | 15 | 15 | 15
Completed | 12 | 14 | 12
Not Completed | 3 | 1 | 3
Not completed — Technical problems/data loss | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anodal TDCS | Cathodal TDCS | Sham TDCS | Total
Number analyzed (Participants) | 12 | 14 | 12 | 38
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.5 (8.06) | 32.4 (14.05) | 32.5 (11.29) | 30.57 (11.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 6 | 8 | 19
  Male | 7 | 8 | 4 | 19

OUTCOME MEASURES:

1. Primary Outcome: Verbal Memory
Description: The Wechsler Memory Scale (WMS-III) is a neuropsychological test designed to measure different memory functions. The WMS-III Word Lists is a measure of verbal learning ability. The examiner reads a list of 12 semantically unrelated words and the subject immediately recalls as many words as possible. For this study, the primary outcome is a measure of verbal recall performance at 24 hours following presentation of the words under three conditions, i.e., anodal tDCS, cathodal tDCS, and sham. Scores may range from 0 (no words recalled) to 12 (all words recalled).
Time Frame: 24 hours
Population: All subjects in this group for whom data were obtained were analyzed
Measure: Mean (Standard Deviation); unit: Words recalled
Groups:
- Left Prefrontal Anodal TDCS: Randomly selected healthy volunteers undergoing left dorsolateral prefrontal cortex (LDPFC) anodal transcranial direct current stimulation (tDCS) during verbal memory tasks.
- Left Prefrontal Cathodal TDCS: Randomly selected healthy volunteers undergoing left dorsolateral prefrontal cortex (LDPFC) cathodal transcranial direct current stimulation (tDCS) during verbal memory tasks.
Arm/Group | Left Prefrontal Anodal TDCS | Left Prefrontal Cathodal TDCS | Sham TDCS
Number analyzed (Participants) | 12 | 14 | 12
Words recalled | 8.625 (1.768) | 9 (1.604) | 8 (2.828)
Statistical Analysis 1: Comparison: Left Prefrontal Anodal TDCS vs Left Prefrontal Cathodal TDCS vs Sham TDCS; Power analysis was based on WMS-III Word Lists performance. With an effect comparable to the effect on verbal fluency in an earlier study of left frontal TDCS in healthy subjects, it would require 10 subjects per group (30 total) for a significance level of 0.05 and 80% power; Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Anodal TDCS | Cathodal TDCS | Sham TDCS
Serious Adverse Events (participants affected / at risk) | 1/12 | 0/14 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/14 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Anodal TDCS (N=12) | Cathodal TDCS (N=14) | Sham TDCS (N=12)
Burn (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) — Punctate burn under reference electrode on arm

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes